CLINICAL TRIAL: NCT06164496
Title: Evaluating the Effectiveness of Different Toothbrushes in Children
Brief Title: Evaluation of the Effectiveness of Different Toothbrushes in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 27.11.2023
Record Dates: First submitted 2023-12-02; First posted 2023-12-11 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Dental Plaque; Plaque, Dental; Oral Hygiene; Gingivitis; Periodontal Indexes
MeSH Terms: conditions — Dental Plaque; Gingivitis

STUDY DESIGN:
Intervention Model Description: single blinded randomized control trial
Who Masked: Investigator
Masking Description: The dental investigator who performed the oral health assessment for dentition status and plaque status was blinded during the intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Experimental): A control group will be formed using a manual brush with a classic head.
  Interventions: Device: standart manual toothbrush
- study group (Experimental): A study group will be formed using a 360-degree bristle brush.
  Interventions: Device: 360 degree toothbrush

INTERVENTIONS:
Device: standart manual toothbrush — Device on plaque removal efficacy
  Arms: control group
Device: 360 degree toothbrush — Device on plaque removal efficacy
  Arms: study group

SUMMARY:
Control groups will be formed in the 2-12 age group using standard manual toothbrushes, and the effectiveness of 360-degree bristle toothbrushes will be compared.

Study design: Experimental study

DETAILED DESCRIPTION:
In this randomized controlled, single-brushing study, children were assigned to a treatment sequence involving a 360-degree toothbrush and a control brush.

Subjects were randomly assigned to a treatment sequence involving a 360-degree toothbrush and a classical manual control toothbrush. Parents brushed the teeth of their children aged 2-5 years, whereas children aged 6-12 years brushed their own teeth under the supervision of clinic staff, unaided by a mirror. Clinical examination of each participant was carried out by the principal investigator. Assessments were done pre- and post-brushing using the "Silness and Löe Plaque Index" (PI), Gingival Index (GI), and the Simplified Oral Hygiene Index (OHI-S). Plaque indices were expressed as means and standard deviations (SD). Within each toothbrush group, the follow-up scores were analyzed using a paired t-test. p < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children aged 2-12.
* Children without systemic disease or developmental dental anomalies.
* Children not undergoing orthodontic treatment.
* Children with no decay on the labial surfaces of upper anterior incisors.
* Patients or their parents accepting participation in the treatment.

Exclusion Criteria:

* Children with decay on the labial surfaces of upper anterior incisors.
* Children undergoing orthodontic treatment.
* Children who, along with their parents, do not agree to participate in the treatment will be excluded from the study.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2023-12-20 (Estimated); Study Completion 2024-01-20 (Estimated)

PRIMARY OUTCOMES:
Within-Treatment Whole-Mouth Differences (vs Baseline) - Plaque removal | 2 weeks
  Mean Change from baseline (pre-brushing to post-brushing) in plaque score after single supervised use based on all surfaces of the whole mouth measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Maltepe, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes